CLINICAL TRIAL: NCT02295228
Title: Hip Arthroplasty and Vitamin D Status
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-1025
Record Dates: First submitted 2014-10-02; First posted 2014-11-20 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D, Vitamin D deficiency, Hip Arthroplasty
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples will be collected at all time points. Blood and urine aliquots will also be banked from each visit.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults undergoing total hip arthroplasty: No intervention will be administered, this is an observational trial. The study population includes adults 50+ who are undergoing elective total hip arthroplasty for osteoarthritis.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There are no interventions. This is an observational trial.

SUMMARY:
It is essential that serum 25(OH)D changes following surgery be clarified, and the mechanism(s) underpinning these changes be identified. As such, the overarching hypothesis of this study is that elective total hip arthroplasty reduces serum total 25(OH)D.

ELIGIBILITY:
Inclusion Criteria:

* Elective total hip arthroplasty for osteoarthritis
* Age 50+
* Able and willing to sign informed consent
* English speaking
* Willing to not alter vitamin D supplementation use for the duration of this study
* Willing to utilize sunscreen of SPF-15 or higher when sun exposure for more than 15 minutes is expected

Exclusion Criteria:

* Illnesses known to affect inflammatory marker status including, but not limited to, rheumatoid arthritis, systemic lupus erythematosis and mixed connective tissue disease
* Chronic diseases that could potentially affect DBP status, e.g., chronic kidney disease stage requiring dialysis, nephrotic syndrome and chronic hepatitis,
* Hip arthritis from causes other than osteoarthritis
* Treatment with medications with potential to affect vitamin D metabolism, (e.g., phenytoin, phenobarbital, teriparatide or active vitamin D analogues) or to potentially interfere with 25(OH)D measurement by HPLC (atavaquone) within the preceding three months.
* Treatment with high dose vitamin D supplementation (50,000 IU weekly or more frequently) within the preceding three months. Note; subjects on a stable daily vitamin D dose will be allowed to participate
* Surgical procedure within the preceding six months
* Use of tanning beds or salons or unwillingness to utilize sunscreen during periods of sun exposure of 15 minutes or longer

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults age 50+ undergoing elective total hip arthroplasty for osteoarthritis will be included. We will exclude individuals having these procedures for other conditions, e.g., rheumatoid arthritis, avascular necrosis and those undergoing reoperation of a previous hip arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in total 25(OH)D | Measured at the pre-operative visit on the day of surgery, post-operative visit (on average 1 to 2 days after surgery), and 6 weeks post-operative visit

SECONDARY OUTCOMES:
DBP (vitamin D binding protein) in serum and urine will be evaluated for 25(OH)D degradation after surgical intervention. | Samples are collected at pre-operative visit on the day of surgery, post-operative (on average 1 to 2 days after surgery) and 6 weeks post-operative visits
  We will evaluate if free 25(OH)D varies over the peri-operative time period. We will evaluate whether the total 25(OH)D change is related to reduced serum DBP and/or increased urinary DBP excretion. We will also correlate the change in free 25(OH)D with serum DBP changes.
Effects of hip arthroplasty on vitamin D metabolite levels in the blood. | Samples are collected at pre-operative visit on the day of surgery, post-operative (on average 1 to 2 days after surgery) and 6 weeks post-operative visits
  We will evaluate the acute and chronic effects of hip arthroplasty on vitamin D metabolites, vitamin D pathway constituents, inflammation, oxidative stress and metabolic markers in plasma using mass spectrometric proteomic and metabolomics analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Binkley, M.D., Principal Investigator — University of Wisconsin, Madison